CLINICAL TRIAL: NCT00566631
Title: Tolerability, Safety and Treatment Response of Flexible Doses of Paliperidone ER in Acutely Exacerbated Subjects With Schizophrenia
Brief Title: An Efficacy and Safety Study of Paliperidone Extended-Release (ER) Tablets in Participants With Schizophrenia
Acronym: PERTAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013162; R076477SCH3018
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Results first posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone Extended Release (ER); Invega
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone Extended Release (ER) (Experimental)
  Interventions: Drug: Paliperidone

INTERVENTIONS:
Drug: Paliperidone — Paliperidone ER tablet in flexible daily dose of 3, 6, 9 or 12 milligram (mg) as per Investigators' discretion will be given once daily orally for 6 weeks in the core treatment phase and no longer than 12 months in the extension phase after the completion of core treatment phase.
  Other Names: Invega

SUMMARY:
The purpose of this study is to evaluate the tolerability, safety and treatment response of flexible doses of paliperidone extended-release (ER; designed to slowly release a drug in the body over an extended period of time) tablets in participants with acute schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-arm (getting one dose of medicine), multi-center (conducted in more than 1 center) study to evaluate tolerability, safety and efficacy of flexible daily doses of paliperidone ER in participants with acute schizophrenia. All participants will be given paliperidone ER once daily at a dose of 3, 6, 9, or 12 milligram (mg) tablets orally depending on Investigator's discretion, based on participant's clinical response and tolerability towards paliperidone ER. The duration of the core phase of the treatment will be 6 weeks and the participants who will complete this phase, respond well and would like to continue, will be eligible to be enrolled in an extension phase, which is no longer than 12 months. Efficacy will primarily be evaluated by treatment response evaluated through total Positive and Negative Syndrome Scale (PANSS) score. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Meets the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria for schizophrenia
* Must be experiencing an acute schizophrenic episode with a Positive and Negative Syndrome Scale (PANSS) total score of greater than or equal to 70 at Baseline
* Must be admitted to hospital for treatment of the acute schizophrenic episode and must agree for voluntary hospitalization for at least the first 7 days of the study
* Female participants must be postmenopausal (for at least 1 year), surgically sterile, abstinent, or, if sexually active, be practicing and effective method of birth control (example, prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study and female participants of child-bearing potential must have a negative urine pregnancy test at Screening
* Participants or their legally acceptable representatives must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Pregnant or breast-feeding female participants
* First antipsychotic treatment ever
* Have received an experimental drug or used an experimental medical device within 30 days before the planned start of treatment and on clozapine or a long-acting injectable antipsychotic during the last 3 months
* Known hypersensitivity to paliperidone extended-release (ER) or risperidone
* Relevant history of any significant or unstable cardiovascular, respiratory, neurologic (including seizures or significant cerebrovascular), renal, hepatic, endocrine, or immunologic diseases, history or current symptoms of tardive dyskinesia or neuroleptic malignant syndrome including recent or present clinically relevant laboratory abnormalities (as deemed by the Investigator) and participants with current or known history (over the past 6 months) of substance dependence according to DSM-IV Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV, Belgium Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (30):
- Zagreb, Croatia
- France (3):
  - Dieppe
  - La Charité-sur-Loire
  - Metz
- Germany (7):
  - Augsburg
  - Bonn
  - Mainz
  - Mannheim
  - München
  - Rostock
  - Wasserburg
- Israel (5):
  - Be-Er Ya-Acov
  - Beersheba
  - Hod HaSharon
  - Pardesiyya
  - Ramat Gan
- Lithuania (3):
  - Klaipėda
  - Šiauliai
  - Vilnius
- Poland (8):
  - Gda Sk Poland
  - Gmina Świecie
  - Lodz
  - Lublin
  - Lubliniec
  - Skąpe
  - Torun
  - Ząbki
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Craiova

REFERENCES:
- See also: Tolerability, Safety and Treatment Response of Flexible Doses of Paliperidone ER in Acutely Exacerbated Subjects With Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=222&filename=CR013162_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone Extended Release (ER): Paliperidone ER tablet in flexible daily dose of 3, 6, 9 or 12 milligram (mg) as per Investigators' discretion was given once daily orally for 6 weeks in the core treatment phase and no longer than 12 months in the extension phase after the completion of core treatment phase.
Period: Part 1: Core Treatment Phase
Arm/Group | Paliperidone Extended Release (ER)
Started | 294
Completed | 234
Not Completed | 60
Not completed — Lack of Efficacy | 18
Not completed — Physician Decision | 1
Not completed — Adverse Event | 9
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 26
Not completed — Moved to a penitentiary hospital | 1
Not completed — Met exclusion criteria | 1
Period: Between Treatment and Extension Phase
Arm/Group | Paliperidone Extended Release (ER)
Started | 234
Completed | 139
Not Completed | 95
Not completed — Participants not willing to participate | 95
Period: Part 2: Extension Phase
Arm/Group | Paliperidone Extended Release (ER)
Started | 139
Completed | 57
Not Completed | 82
Not completed — Lack of Efficacy | 25
Not completed — Withdrawal by Subject | 34
Not completed — Adverse Event | 11
Not completed — Lost to Follow-up | 6
Not completed — Death | 1
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 294
Age Continuous [Mean (Standard Deviation); unit: Years] | 40.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138
  Male | 156

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Response Based on Total PANSS Scale Score
Description: Response was defined as decrease of at least 30 percent in total Positive and Negative Syndrome Scale (PANSS) score from Baseline to endpoint of core phase (which is, Day 42 or early discontinuation). The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, & poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of sum of all 30 PANSS items & ranges from 30 to 210. Higher scores indicate worsening.
Time Frame: Day 42 or early discontinuation
Population: Intent-to-treat (ITT) population included all participants who received at least one dose of paliperidone ER and provided at least 1 post-baseline efficacy measurement.
Measure: Number; unit: Participants
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 294
Participants | 195

2. Secondary Outcome: Change From Baseline in Total Positive and Negative Symptom Scale (PANSS) Score at Day 2, 3, 4, 5, 7, 14, 28, 42 and Final Evaluation (Day 42 or Early Discontinuation)
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening. Final evaluation is the last post-baseline visit with data.
Time Frame: Baseline, Day 2, 3, 4, 5, 7, 14, 28, 42 and Final Evaluation (Day 42 or early discontinuation)
Population: The ITT population included all participants who received at least one dose of paliperidone ER and provided at least 1 post-baseline efficacy measurement. "n" signifies those participants who were evaluated for this measure at given time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 294
Units on a scale
  Baseline (n=294) | 100.2 (17.2)
  Change at Day 2 (n=294) | -2.3 (5.3)
  Change at Day 3 (n=287) | -5.8 (7.9)
  Change at Day 4 (n=288) | -10.3 (11.3)
  Change at Day 5 (n=284) | -13.3 (13.3)
  Change at Day 7 (n=286) | -17.4 (15.5)
  Change at Day 14 (n=276) | -22.3 (16.0)
  Change at Day 28 (n=254) | -27.2 (16.6)
  Change at Day 42 (n=234) | -32.1 (17.5)
  Change at Final Evaluation (n=294) | -27.5 (20.1)

3. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Marder Subscale Scores at Day 42 and Final Evaluation (Day 42 or Early Discontinuation)
Description: The PANSS is a 30-item scale to assess neuropsychiatric symptoms of schizophrenia. The symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme psychopathology). Positive symptoms subscale consists of 8 items with total score range of 8-56; negative symptoms and disorganized thoughts subscale, consists of 7 items with total score range of 7-49, uncontrolled hostility/excitement (H/E) subscale and anxiety/depression subscale, each consists of 4 items with total score range of 4-28. Higher score indicates greater severity. Final evaluation is the last post-baseline visit with data.
Time Frame: Baseline, Day 42 and Final Evaluation (Day 42 or early discontinuation)
Population: The ITT population included all participants who received at least one dose of paliperidone ER and provided at least 1 post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 294
Units on a scale
  Positive Score: Baseline | 28.8 (5.8)
  Positive Score: Change at Day 42 | -10.6 (5.9)
  Positive Score: Change at Final Evaluation | -9.1 (6.7)
  Negative Score: Baseline | 24.8 (6.1)
  Negative Score: Change at Day 42 | -6.5 (5.1)
  Negative Score: Change at Final Evaluation | -5.7 (5.3)
  Disorganized Thoughts: Baseline | 23.4 (4.9)
  Disorganized Thoughts: Change at Day 42 | -6.5 (4.6)
  Disorganized Thoughts: Change at Final Evaluation | -5.6 (5.0)
  Uncontrolled H/E: Baseline | 10.6 (3.7)
  Uncontrolled H/E: Change at Day 42 | -3.8 (3.2)
  Uncontrolled H/E: Change at Final Evaluation | -3.2 (3.8)
  Anxiety/Depression: Baseline | 12.5 (3.2)
  Anxiety/Depression: Change at Day 42 | -4.8 (3.2)
  Anxiety/Depression: Change at Final Evaluation | -3.9 (3.7)

4. Secondary Outcome: Percentage of Participants With Treatment Response Greater Than (>) 20 Percent, 40 Percent and 50 Percent in Total Positive and Negative Syndrome Scale (PANSS) Score
Description: as for outcome 2
Time Frame: Day 2, 3, 4, 5, 7, 14, 28, 42 and Final Evaluation (Day 42 or early discontinuation)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 294
Percentage of participants
  Treatment Response>20 Percent at Day 2 | 4.4
  Treatment Response>20 Percent at Day 3 | 12.9
  Treatment Response>20 Percent at Day 4 | 29.9
  Treatment Response>20 percent at Day 5 | 39.4
  Treatment Response>20 Percent at Day 7 | 55.6
  Treatment Response>20 Percent at Day 14 | 72.1
  Treatment Response>20 Percent at Day 28 | 79.9
  Treatment Response>20 percent at Day 42 | 87.6
  Treatment Response>20 Percent at Final Evaluation | 76.5
  Treatment Response>40 Percent at Day 2 | 0
  Treatment Response>40 Percent at Day 3 | 1.7
  Treatment Response>40 Percent at Day 4 | 6.9
  Treatment Response>40 Percent at Day 5 | 11.6
  Treatment Response>40 Percent at Day 7 | 19.6
  Treatment Response>40 Percent at Day 14 | 33.7
  Treatment Response>40 Percent at Day 28 | 48.0
  Treatment Response>40 Percent at Day 42 | 59.4
  Treatment Response>40 Percent at Final Evaluation | 51.4
  Treatment Response>50 Percent at Day 2 | 0
  Treatment Response>50 Percent at Day 3 | 0
  Treatment Response>50 Percent at Day 4 | 2.8
  Treatment Response>50 Percent at Day 5 | 7.4
  Treatment Response>50 Percent at Day 7 | 11.2
  Treatment Response>50 Percent at Day 14 | 18.1
  Treatment Response>50 Percent at Day 28 | 29.9
  Treatment Response>50 Percent at Day 42 | 41.5
  Treatment Response>50 Percent at Final Evaluation | 34.7

5. Secondary Outcome: Change From Baseline in Clinical Global Impression -Severity (CGI-S) Score at Day 7, 14, 28, 42 and Final Evaluation (Day 42 or Early Discontinuation)
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "normal, not at all ill" and a rating of 7 is equivalent to "among the most extremely ill participants". Higher scores indicate worsening. Final evaluation is the last post-baseline visit with data.
Time Frame: Baseline, Day 7, 14, 28, 42 and Final Evaluation (Day 42 or early discontinuation)
Population: The ITT population included all participants who received at least 1 dose of paliperidone ER and provided at least 1 post-baseline efficacy measurement. "N" (number of participants analyzed) signifies those participants who were evaluable for this measure and "n" signifies those participants who were evaluated for this measure at given time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 289
Units on a scale
  Baseline (n=289) | 3.9 (0.7)
  Change at Day 7 (n=286) | -0.6 (0.7)
  Change at Day 14 (n=275) | -0.9 (0.8)
  Change at Day 28 (n=253) | -1.2 (0.9)
  Change at Day 42 (n=234) | -1.5 (0.9)
  Change at Final Evaluation (n=289) | -1.2 (1.0)

6. Secondary Outcome: Change From Baseline in Personal and Social Performance Scale (PSP) Score at Day 7, 14, 28, 42 and Final Evaluation (Day 42 or Early Discontinuation)
Description: The PSP assesses the degree of dysfunction within 4 domains of behavior: socially useful activities, personal & social relationships, self-care & disturbing and aggressive behavior. The score ranges from 1 to 100, divided into 10 equal intervals to rate the degree of difficulty (1, absent to 6, very severe) in each of 4 domains. Participants with a score of 71 to 100 have a mild degree of difficulty; from 31 to 70, varying degrees of disability; less than or equal to 30, functioning so poorly as to require intensive supervision. Final evaluation is the last post-baseline visit with data.
Time Frame: Baseline, Day 7, 14, 28, 42 and Final Evaluation (Day 42 or early discontinuation)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 290
Units on a Scale
  Baseline (n=290) | 50.0 (14.3)
  Change at Day 7 (n=287) | 6.3 (9.5)
  Change at Day 14 (n=276) | 9.9 (10.5)
  Change at Day 28 (n=254) | 13.8 (12.3)
  Change at Day 42 (n=235) | 16.1 (13.9)
  Change at Final Evaluation (n=290) | 13.7 (14.4)

7. Secondary Outcome: Change From Baseline in Quality of Sleep Evaluation Score at Day 7, 14, 28, 42 and Final Evaluation (Day 42 or Early Discontinuation)
Description: The sleep evaluation scale is a self-administered scale that rates quality of sleep. Participants indicate on an 11-point scale that how well they have slept within the previous 7 days, score ranged from 0 (very badly) to 10 (very well). Final evaluation is the last post-baseline visit with data.
Time Frame: Baseline, Day 7, 14, 28, 42 and Final Evaluation (Day 42 or early discontinuation)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 286
Units on a scale
  Baseline (n=286) | 5.4 (2.8)
  Change at Day 7 (n=280) | 1.4 (2.9)
  Change at Day 14 (n=273) | 1.7 (2.9)
  Change at Day 28 (n=250) | 2.1 (3.0)
  Change at Day 42 (n=234) | 2.6 (2.9)
  Change at Final Evaluation (n=286) | 2.1 (3.2)

8. Secondary Outcome: Change From Baseline in Day Time Drowsiness Evaluation Score at Day 7, 14, 28, 42 and Final Evaluation (Day 42 or Early Discontinuation)
Description: The day time drowsiness evaluation scale is a self-administered scale that rates day time drowsiness. Participants indicate on an 11-point scale that how often they have felt drowsy within the previous 7 days, score ranged from 0 (not at all) to 10 (all the time). Final evaluation is the last post-baseline visit with data.
Time Frame: Baseline, Day 7, 14, 28, 42 and Final Evaluation (Day 42 or early discontinuation)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 286
Units on a scale
  Baseline (n=286) | 3.4 (2.7)
  Change at Day 7 (n=280) | -0.5 (2.5)
  Change at Day 14 (n=273) | -1.0 (2.6)
  Change at Day 28 (n=250) | -1.4 (2.7)
  Change at Day 42 (n=234) | -1.6 (2.6)
  Change at Final Evaluation (n=286) | -1.4 (2.7)

9. Secondary Outcome: Number of Participants Satisfied With the Study Treatment
Description: Treatment satisfaction with paliperidone ER was assessed by the Investigator and participant on a 5-point scale: 1 (very good), 2 (good), 3 (reasonable), 4 (moderate) and 5 (poor), at the end of the core treatment phase (which is, Day 42 or early discontinuation) by conducting an interview.
Time Frame: Day 42 or early discontinuation
Population: The ITT population included all participants who received at least 1 dose of paliperidone ER and provided at least 1 post-baseline efficacy measurement. "N" (number of participants analyzed) signifies those participants who were evaluable for this measure at given time point.
Measure: Number; unit: Participants
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 268
Participants
  Treatment efficacy: Very good | 66
  Treatment efficacy: Good | 111
  Treatment efficacy: Reasonable | 53
  Treatment efficacy: Moderate | 25
  Treatment efficacy: Poor | 13
  Treatment tolerability: Very good | 84
  Treatment tolerability: Good | 124
  Treatment tolerability: Reasonable | 35
  Treatment tolerability: Moderate | 15
  Treatment tolerability: Poor | 10

10. Other Pre Specified Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Score at Day 7, 14, 42 and Final Evaluation (Day 42 or Early Discontinuation)
Description: The AIMS is a 12-item scale to provide a numeric measure to the observed abnormal movements in different parts of the body. Information is collected after a brief neurological examination and is scored on a 5-point scale (0=none and 4=severe). Final evaluation is the last post-baseline visit with data.
Time Frame: Baseline, Day 7, 14, 42 and Final Evaluation (Day 42 or early discontinuation)
Population: Safety population included all participants who received at least 1 dose of paliperidone ER and had at least 1 post-baseline safety assessment. "N" (number of participants analyzed) signifies those participants who were evaluable for this measure and "n" signifies those participants who were evaluated for this measure at given time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 290
Units on a scale
  Baseline (n=290) | 0.59 (2.0)
  Change at Day 7 (n=287) | -0.05 (1.2)
  Change at Day 14 (n=276) | -0.13 (1.3)
  Change at Day 42 (n=234) | -0.18 (1.7)
  Change at Final Evaluation (n=290) | -0.09 (1.8)

11. Other Pre Specified Outcome: Change From Baseline in Simpson Angus Extrapyramidal Symptoms Rating Scale (SAS) Score at Day 7, 14, 42 and Final Evaluation (Day 42 or Early Discontinuation)
Description: The SAS is a 10-item scale used to measure the symptoms of parkinsonism (slow movements) or parkinsonian side-effects related to the use of antipsychotic medications. The SAS rates 10 items (including gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, leg pendulousness, head dropping, Glabella tap, tremor and salivation), score ranging from 0 (normal) to 4 (extreme). The SAS global score is the average score (total sum of items score divided by the number of items) and ranges between 0 and 4, where the higher score indicates more severe condition of Extrapyramidal Symptoms. Final evaluation is the last post- baseline visit with data.
Time Frame: Baseline, Day 7, 14, 42 and Final Evaluation (Day 42 or early discontinuation)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 290
Units on a scale
  Baseline (n=290) | 0.16 (0.32)
  Change at Day 7 (n=287) | 0.00 (0.23)
  Change at Day 14 (n=276) | -0.00 (0.24)
  Change at Day 42 (n=234) | -0.02 (0.24)
  Change at Final Evaluation (n=290) | 0.01 (0.34)

12. Other Pre Specified Outcome: Change From Baseline in Global Rating Sub-scale Score Based on Barnes Akathisia Rating Scale (BARS) at Day 7, 14, 42 and Final Evaluation (Day 42 or Early Discontinuation)
Description: The BARS included an objective rating (from 0=normal to 3=constantly engaged), two subjective ratings of symptoms of akathisia, namely awareness of restlessness (ranging from 0=absence of inner restlessness to 3=awareness of intense compulsion to move) and reported distress related to restlessness (ranging from 0=no distress to 3=severe), and a global clinical rating of akathisia, ranging from 0 (absent) to 5 (severe). Global rating sub-scale score (that is, global clinical rating of akathisia) was assessed which was scored separately and is the most relevant measure of severity of akathisia. Higher scores indicates worsening akathisia. Final evaluation is the last post-baseline visit with data.
Time Frame: Baseline, Day 7, 14, 42 and Final Evaluation (Day 42 or early discontinuation)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 290
Units on a scale
  Baseline (n=290) | 0.17 (0.5)
  Change at Day 7 (n=286) | -0.02 (0.4)
  Change at Day 14 (n=276) | -0.01 (0.5)
  Change at Day 42 (n=234) | -0.03 (0.5)
  Change at Final Evaluation (n=290) | 0.03 (0.7)

ADVERSE EVENTS:
Time Frame: 6 weeks in the core treatment phase
Description: An adverse event is any untoward medical occurrence in a clinical study participant administered with study treatment. It can be any unfavorable
  & unintended sign/abnormal finding, symptom, or disease temporally associated with use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Arm/Group | Paliperidone Extended Release (ER)
Serious Adverse Events (participants affected / at risk) | 23/294
Other Adverse Events (participants affected / at risk) | 150/294
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Extended Release (ER) (N=294)
Tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Extrapyramidal disorder (Nervous system disorders) | 2
Mental impairment (Nervous system disorders) | 1
Acute psychosis (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Intentional self-injury (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 12
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Extended Release (ER) (N=294)
Tachycardia (Cardiac disorders) | 25
Constipation (Gastrointestinal disorders) | 9
Nasopharyngitis (Infections and infestations) | 13
Akathisia (Nervous system disorders) | 13
Extrapyramidal disorder (Nervous system disorders) | 18
Headache (Nervous system disorders) | 22
Agitation (Psychiatric disorders) | 10
Anxiety (Psychiatric disorders) | 14
Insomnia (Psychiatric disorders) | 68
Restlessness (Psychiatric disorders) | 10
Sleep disorder (Psychiatric disorders) | 9
Hypertension (Vascular disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days